CLINICAL TRIAL: NCT02271048
Title: The Feasibility and Effectiveness Study for Clinical Application of Realtime Tele-ultrasonography Using the Smartphone
Brief Title: The Feasibility and Effectiveness Study for Tele-ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Changsun Kim, Clinical assistant professor, Hanyang University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2014-03
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Teleradiology
Keywords: telemedicine; ultrasonography; echocardiography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): The raters in this group one firstly review ultrasound images numbered from one to 50 using LCD monitor of ultrasound machine and after mandatory rests of 20 minutes, review the remaining ultrasound examinations numbered from 51 to 100 using iPhone display with CubeView at their first visit.(Remote ultrasonography interpretation using the smartphone)
  They visited twice with an interval of four weeks and reviewed the ultrasound images using revered devices at each session.
  Interventions: Device: Remote ultrasonography interpretation using the smartphone
- Group II (Experimental): The raters in this group II firstly review the ultrasound images numbered from one to 50 using iPhone with CubeView (Remote ultrasonography interpretation using the smartphone) and 51 to 100 with the LCD monitor.
  They visited twice with an interval of four weeks and reviewed the ultrasound images using revered devices at each session.
  Interventions: Device: Remote ultrasonography interpretation using the smartphone

INTERVENTIONS:
Device: Remote ultrasonography interpretation using the smartphone — The reviewers interpreted the ultrasonography images on the smartphone transmitted from the ultrasound machine in real time
  Other Names: Smartphone (A1530, iPhone 5S, USA)

SUMMARY:
Purpose

- The investigators aim to evaluate the feasibility of remote interpretation for ultrasound images using a smartphone based realtime image transmission system.

Methods

A total of 100 echocardiography examinations; 50 showed the ejection fraction above 50% and remaining 50 cases showed the ejection fraction under 50%, and 100 abdominal ultrasound images; 50 had signs of acute appendicitis and the other 50 had no findings of appendicitis will be consecutively selected. The 12 raters review these original images using an LCD monitor of the ultrasound machine and also an iPhone which is connected to the ultrasound machine via remote image transmission system (CubeView, Alpinion medical system, Seoul, Korea), evaluating left ventricular systolic function (for echocardiography) by measuring the ejection fraction and grading the probability of presence of acute appendicitis on each examination by a five Likert scale.

The sensitivity and specificity between two devices will be compared and the diagnostic performance between two devices will be also compared. The image quality between two devices will be measured using the double stimulation impairment scale (DSIS)

DETAILED DESCRIPTION:
The 12 raters are randomly divided into two groups

The raters in group one review the echocardiographies examinations numbered from one to 50 using LCD monitor of ultrasound machine and review the remaining 50 examinations numbered from 51 to 100 using iPhone with CubeView at their first visit The other group firstly review echocardiography numbered from one to 50 using iPhone with CubeView and 51 to 100 with the LCD monitor.

They visit twice with an interval of four weeks and review the echocardiography examinations using revered devices at each session. They also review abdominal ultrasound images on the same plan as reviewing echocardiography.

When they review the echocardiography, the raters measure the ejection fraction by visual estimation (1=obviously normal EF, 2 = probably normal EF, 3 = unsure, 4 = probably reduced EF, 5 = obviously reduced EF). In cate of d the abdominal ultrasound, they are instructed to rate the likelihood of the presence or absence of appendicitis in each case using a five-Likert scale (1 = obvious no appendicitis, 2 = unlikely appendicitis, 3 = unsure, 4 = likely appendicitis, 5 = obvious appendicitis).

ELIGIBILITY:
Inclusion Criteria:

* Board certified emergency physicians with a ultrasound experience of 4 years and over.

Exclusion Criteria:

* Corrected eyesight < 20/30
* Color weakness or blindness

Ages: 33 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance between iPhone and LCD monitor | within one day
  Dorfman-Berbaum-Metz method with RSCORE and semi-parametric estimation of ROC indices by using the DMB-MRMC software (version 2.3, available at http://perception.radiology.uiowa.edu)
  * 95% confidence interval
  * The reviewers and cases are taken as random factors

CONTACTS AND LOCATIONS:
Overall Officials: Bo Seung Kang, MD, Study Director — Hanyang University Guri Hospital
Locations (1):
- Hanyang university guri hospital, Department of emergency medicine, Guri-si, GyeongGido, South Korea

REFERENCES:
- [Background] Adambounou K, Farin F, Boucher A, Adjenou KV, Gbeassor M, N'dakena K, Vincent N, Arbeille P. [System of telesonography with synchronous teleconsultations and asynchronous telediagnoses (Togo)]. Med Sante Trop. 2012 Jan-Mar;22(1):54-60. doi: 10.1684/mst.2012.0002. French. PMID 22868727
- [Background] Sable CA, Cummings SD, Pearson GD, Schratz LM, Cross RC, Quivers ES, Rudra H, Martin GR. Impact of telemedicine on the practice of pediatric cardiology in community hospitals. Pediatrics. 2002 Jan;109(1):E3. doi: 10.1542/peds.109.1.e3. PMID 11773571
- [Background] Costa C, Oliveira JL. Telecardiology through ubiquitous internet services. Int J Med Inform. 2012 Sep;81(9):612-21. doi: 10.1016/j.ijmedinf.2012.05.011. Epub 2012 Jun 17. PMID 22709977
- [Background] Paulus YM, Thompson NP. Inexpensive, realtime tele-ultrasound using a commercial, web-based video streaming device. J Telemed Telecare. 2012 Jun;18(4):185-8. doi: 10.1258/jtt.2012.110112. Epub 2012 May 25. PMID 22637653
- [Background] Ogedegbe C, Morchel H, Hazelwood V, Chaplin WF, Feldman J. Development and evaluation of a novel, real time mobile telesonography system in management of patients with abdominal trauma: study protocol. BMC Emerg Med. 2012 Dec 18;12:19. doi: 10.1186/1471-227X-12-19. PMID 23249290
- [Background] McBeth P, Crawford I, Tiruta C, Xiao Z, Zhu GQ, Shuster M, Sewell L, Panebianco N, Lautner D, Nicolaou S, Ball CG, Blaivas M, Dente CJ, Wyrzykowski AD, Kirkpatrick AW. Help is in your pocket: the potential accuracy of smartphone- and laptop-based remotely guided resuscitative telesonography. Telemed J E Health. 2013 Dec;19(12):924-30. doi: 10.1089/tmj.2013.0034. Epub 2013 Oct 19. PMID 24138615
- [Background] Biegler N, McBeth PB, Tiruta C, Hamilton DR, Xiao Z, Crawford I, Tevez-Molina M, Miletic N, Ball CG, Pian L, Kirkpatrick AW. The feasibility of nurse practitioner-performed, telementored lung telesonography with remote physician guidance - 'a remote virtual mentor'. Crit Ultrasound J. 2013 Jun 27;5(1):5. doi: 10.1186/2036-7902-5-5. PMID 23805869
- [Derived] Kim C, Cha H, Kang BS, Choi HJ, Lim TH, Oh J. A Feasibility Study of Smartphone-Based Telesonography for Evaluating Cardiac Dynamic Function and Diagnosing Acute Appendicitis with Control of the Image Quality of the Transmitted Videos. J Digit Imaging. 2016 Jun;29(3):347-56. doi: 10.1007/s10278-015-9849-6. PMID 26620200